CLINICAL TRIAL: NCT00969644
Title: The Relationship Between the Growth Hormone (GH)- Insulin Like Growth Factor I (IGF-I) System and the Inflammatory System in Healthy Normal Persons
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Herlev Hospital (Other)
Responsible Party: Mikkel Andreassen, MD., Department of Endocrinology, Herlev Hospital, 2730 Herlev Ringvej 75, Herlev
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: HC-2009-049
Record Dates: First submitted 2009-08-31; First posted 2009-09-01 (Estimated); Last update posted 2009-09-01 (Estimated); Status verified 2009-08

CONDITIONS: Interaction Between the GH/IGF-I System and the Immune-system
MeSH Terms: interventions — Human Growth Hormone; pegvisomant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GH (Active Comparator)
  Interventions: Drug: Somatropin
- Pegvisomant (Active Comparator)
  Interventions: Drug: Pegvisomant

INTERVENTIONS:
Drug: Somatropin — s.c injections once daily 10-30 mícrogram/kg/day
  Arms: GH
Drug: Pegvisomant — s.c. injections once daily (10-15 mg/day)
  Arms: Pegvisomant

SUMMARY:
Observations in patients with growth hormone (GH)-disturbances have suggested that GH/IGF-I might have anti-inflammatory effects. To elucidate this hypothesis the investigators have planned a study to investigate if 3 weeks administration of GH and subsequently the GH antagonist Pegvisomant (or vice versa) influence serum levels of different inflammatory markers in healthy volunteers.

DETAILED DESCRIPTION:
To investigate if administration of 3 weeks og GH (10-30 microgram/kg/day) and subsequent Pegvisomant (10-15 mg/day) influence serum concentrations of the inflammatory variables Tumor Necrosis Factor α (TNF-α), Interleukin-6 (IL-6), high sensitive CRP (hsCRP) and the newly discovered acute phase protein YKL-40. The study involves 12 healthy volunteers age from 22-65 years.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, normal blood tests

Exclusion Criteria:

* Previous cancer

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2009-09; Primary Completion 2010-03 (Estimated); Study Completion 2010-03 (Estimated)

PRIMARY OUTCOMES:
The relationship between changes in serum levels of Tumor Necrosis Factor α (TNF-α), Interleukin-6 (IL-6), high sensitive CRP (hsCRP) and YKL-40 vs. changes in serum levels og IGF-I | 1/9 2009 - 1/3 2010

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Endocrinology J 106, Herlev Hospital, Herlev, Herlev, Denmark

REFERENCES:
- [Derived] Andreassen M, Frystyk J, Faber J, Kristensen LO, Juul A. Growth hormone (GH) activity is associated with increased serum oestradiol and reduced anti-Mullerian hormone in healthy male volunteers treated with GH and a GH antagonist. Andrology. 2013 Jul;1(4):595-601. doi: 10.1111/j.2047-2927.2013.00096.x. PMID 23785020